CLINICAL TRIAL: NCT05533684
Title: A Single Preoperative Dose of Gabapentin to Decreases Postoperative Pain in Ambulatory Anal Surgeries
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Sarah Mohamed Aly Omar Mousa, principal investigator, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 343-2022
Record Dates: First submitted 2022-09-03; First posted 2022-09-09 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Pain, Postoperative
Keywords: anal surgery,; gabapentin,; postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Gabapentin

STUDY DESIGN:
Intervention Model Description: 2 groups are included in the study
Who Masked: Participant, Investigator
Masking Description: double-blinded study both participant and investigator are blind to the study drug
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- postoperative pain (No Intervention): Measuring postoperative pain using the visual analogue scale
- total analgesic consumption (Other): Recording the total amount of analgesia consumed by the patients
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Gabapentin — single preoperative dose of 600 mg gabapentin
  Other Names: Gaptin 600 mg
  Arms: total analgesic consumption

SUMMARY:
Single dose 600 mg gabapentin will be given preoperatively in anal surgeries

DETAILED DESCRIPTION:
Patients will be grouped into 2 groups of 25 patients each, the first group will receive 600 mg of gabapentin one hour before surgery and the second group will receive a placebo tablet. pain scores will be measured postoperatively

ELIGIBILITY:
Inclusion Criteria:

1. ASA physical status I or II
2. Aged from 18 to 65 years
3. Scheduled for anal surgeries at Minya University Hospital

Exclusion Criteria:

1. Presence of contraindications to neuraxial anesthesia
2. Presence of history of central nervous system or mental disorders, epilepsy, chronic pain, or drug abuse.
3. The use of neuropathic analgesic or antiepileptic drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
postoperative pain | first 12 hours postoperative
  measuring postoperative pain using the visual analog scale from 0 to 10, where zero is the least, and 10 is the worst pain

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Omar, M.D., Principal Investigator — Minia University
Locations (1):
- Sarah Omar, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No
The research will be available to other researchers when it is completed